CLINICAL TRIAL: NCT03087292
Title: Effect of Low Intensity Resistance Training With Vascular Occlusion on Muscle Hypertrophy, Neuromuscular Adaptations and Selected Cardiovascular Parameters in Patients With Coronary Heart Disease
Brief Title: Low Intensity Resistance Training With Vascular Occlusion in Coronary Heart Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Assistant Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLRehab022017
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Coronary Disease; Coronary Artery Disease
Keywords: blood flow restriction; resistance training; coronary heart disease
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training group (Active Comparator): Patients to be randomly assigned to the "resistance training group" will have resistance training with vascular occlusion 2 times per week for a period of 8 weeks on unilateral leg extension machine. During each training, they will performed 3 sets of 15 repetitions at the intensity of 30% 1 RM (repetition maximum). Each training set will separated by a 30 second rest period.
  Interventions: Other: Resistance training with vascular occlusion
- Control group (No Intervention): Patients to be randomly assigned to the control group (normal physical activity) will continue with their usual physical activity regime.

INTERVENTIONS:
Other: Resistance training with vascular occlusion — Patients will perform unilateral leg extension resistance training with vascular occlusion 2 times per week for a period of 8 weeks. Each training session will consist of 3 sets of 15 repetitions at the intensity of 30% 1 RM with 30 s of rest period between sets.
  Arms: Resistance training group

SUMMARY:
In our clinical controlled trial, patients with coronary heart disease will be randomly assigned into the exercise intervention (low intensity resistance training with vascular occlusion) or usual physical activity group (control group).

DETAILED DESCRIPTION:
Physical activity in patients with coronary heart disease improves health, quality of life, and reduces risk of coronary events, morbidity and mortality. Aerobic training is preferred as a part of cardiac rehabilitation with its well established evidence-based guidelines. On the other hand, the resistance training was first introduced as a part of cardiac rehabilitation just over a decade ago, due to its positive effects on performance, quality of life and muscle hypertrophy and strength. Despite the positive effects of resistance training, there still lacks evidence about its effect on cardiovascular health. Furthermore, guidelines still do not specify the exact training volumes, doses and types of resistance training for patients with coronary heart disease.

In clinical practice, it is often difficult and contraindicated to use near-maximal loads (e.g., in the early stages of cardiac rehabilitation, after sport injury, etc.). Muscle atrophy and weakness often occur rapidly in the affected area due to the effects of trauma (or disease) and inactivity. Consequently, training modalities that promote hypertrophy or counteract atrophy without the use of heavy loads should be of special interest in the rehabilitation of some chronic diseases for which high musculoskeletal forces are contraindicated.

Occlusive strength training with tourniquet cuffs was first used nearly twenty years ago. Studies have shown that low to-moderate intensity (20-50% of 1RM) resistance training with vascular occlusion leads to gains in muscle strength and volume comparable to those seen after conventional heavy resistance training. This effects suggest, that ischemic strength training may be a useful method in rehabilitation and other contexts.

To conclude, the aim of this study is to compare the effect of low intensity resistance training with vascular occlusion vs. normal physical activity on:

1. muscle hypertrophy, strength and neuromuscular parameters;
2. vascular function;
3. and blood parameters (anabolic and catabolic hormones, catecholamines, inflammations factors, parameters of oxidative stress etc.)

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old and below 75 years old
* coronary heart disease documented with clinical event
* stable coronary heart disease patients

Exclusion Criteria:

* Unstable phase of coronary heart disease
* dysfunction of left ventricle
* residual myocardial ischemia
* contraindications for physical activity,
* intellectual development disorder,
* recent dissection of aorta
* recent vein thrombolysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-06-15 (Estimated); Study Completion 2017-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in maximal strength | 4 weeks, 8 weeks
  Determined with one repetition maximum test on leg extension machine (kg)

SECONDARY OUTCOMES:
Change in maximal voluntary contraction (MVC) | 4 and 8 weeks
  Determined with modified interpolated twitch protocol
Changes of flow-mediated dilatation of the brachial artery | 4 weeks, 8 weeks
  Measured with ultrasound in %
Change in muscle hypertrophy (muscle thickness) | 4 and 8 weeks
  Measured with ultrasound in mm
Change of the value of blood human growth hormon (HGH) | 4 and 8 weeks
  measured in ng/mL
Change of the value of testosterone | 4 and 8 weeks
  measured in ng/dL
Change of the value of myostatin | 4 and 8 weeks
  measured in ng/mL
Change of the value of mechano growth factor (MGF) | 4 and 8 weeks
  measured in ng/mL
Change of the value of insulin-like growth factor (IGF-1) | 4 and 8 weeks
  measured in ng/mL
Change of the value of epinephrine | 4 and 8 weeks
  measured in pg/mL
Change of the value of norepinephrine | 4 and 8 weeks
  measured in pg/mL
Change of the value of cortisol | 4 and 8 weeks
  measured in mcg/dL
Change in C-reactive protein | 4 and 8 weeks
  measured in mg/L
Change in blood pressure prior and after exercise | 1-8 week
  measured in mmHg
Change in heat-shock protein (HSP-72) | 4 and 8 weeks
  measured in ng/mL
Change in resting and post-exercise heart rate | 4 and 8 weeks
  Measured in beats per min
Change of from-the-questionnaire-obtained quality of life | 4 and 8 weeks
  Measured in points

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

REFERENCES:
- [Background] Nakajima, T., et al. Use and safety of KAATSU training: results of a national survey. Int J KAATSU Train Res; 2(1): 5-13, 2006.
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889
- [Background] Pollock ML, Franklin BA, Balady GJ, Chaitman BL, Fleg JL, Fletcher B, Limacher M, Pina IL, Stein RA, Williams M, Bazzarre T. AHA Science Advisory. Resistance exercise in individuals with and without cardiovascular disease: benefits, rationale, safety, and prescription: An advisory from the Committee on Exercise, Rehabilitation, and Prevention, Council on Clinical Cardiology, American Heart Association; Position paper endorsed by the American College of Sports Medicine. Circulation. 2000 Feb 22;101(7):828-33. doi: 10.1161/01.cir.101.7.828. No abstract available. PMID 10683360
- [Background] Karabulut M, Abe T, Sato Y, Bemben MG. The effects of low-intensity resistance training with vascular restriction on leg muscle strength in older men. Eur J Appl Physiol. 2010 Jan;108(1):147-55. doi: 10.1007/s00421-009-1204-5. Epub 2009 Sep 18. PMID 19760431
- [Background] Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T, Dhanani S, Volpi E, Rasmussen BB. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol (1985). 2010 May;108(5):1199-209. doi: 10.1152/japplphysiol.01266.2009. Epub 2010 Feb 11. PMID 20150565
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Heran BS, Chen JM, Ebrahim S, Moxham T, Oldridge N, Rees K, Thompson DR, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD001800. doi: 10.1002/14651858.CD001800.pub2. PMID 21735386
- [Derived] Kambic T, Novakovic M, Tomazin K, Strojnik V, Bozic-Mijovski M, Jug B. Hemodynamic and Hemostatic Response to Blood Flow Restriction Resistance Exercise in Coronary Artery Disease: A Pilot Randomized Controlled Trial. J Cardiovasc Nurs. 2021 Sep-Oct 01;36(5):507-516. doi: 10.1097/JCN.0000000000000699. PMID 32496365
- [Derived] Kambic T, Novakovic M, Tomazin K, Strojnik V, Jug B. Blood Flow Restriction Resistance Exercise Improves Muscle Strength and Hemodynamics, but Not Vascular Function in Coronary Artery Disease Patients: A Pilot Randomized Controlled Trial. Front Physiol. 2019 Jun 12;10:656. doi: 10.3389/fphys.2019.00656. eCollection 2019. PMID 31244668